CLINICAL TRIAL: NCT00494442
Title: A Phase II Open-label, Non-comparative, International, Multicentre Study to Assess the Efficacy and Safety of KU 0059436 Given Orally Twice Daily in Patients With Advanced BRCA1 or BRCA2 Associated Ovarian Cancer
Brief Title: Study to Assess the Efficacy and Safety of a PARP Inhibitor for the Treatment of BRCA-positive Advanced Ovarian Cancer
Acronym: ICEBERG 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: KuDOS Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU36-58; D0810C00009
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Neoplasm
Keywords: Advanced ovarian cancer; Poly(ADP ribose) polymerases; KU-0059436; AZD2281; BRCA1 protein; BRCA2 protein
MeSH Terms: conditions — Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KU-0059436 (AZD2281) 100 mg BID (Experimental)
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor)
- KU-0059436 (AZD2281) 400 mg BID (Experimental)
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor)

INTERVENTIONS:
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Other Names: Olaparib
  Arms: KU-0059436 (AZD2281) 100 mg BID
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Arms: KU-0059436 (AZD2281) 400 mg BID

SUMMARY:
The purpose of the study is to see if the drug KU 0059436 is effective and well tolerated in treating patients with measurable BRCA1- or BRCA2-positive advanced ovarian cancer and for whom no curative therapeutic option exists.

ELIGIBILITY:
Inclusion Criteria:

* Advanced ovarian cancer with positive BRCA1 or BRCA2 status
* Failed at least one prior chemotherapy
* In investigators opinion, no curative standard therapy exists
* Measurable disease

Exclusion Criteria:

* Brain metastases
* Less than 28 days since last treatment used to treat the disease
* Considered a poor medical risk due to a serious uncontrolled disorder

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-06-11 (Actual); Primary Completion 2009-03-17 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Carmichael, BSc MBChB MD FRCP, Study Director — KuDOS Pharmaceuticals Limited; Andrew Tutt, PhD MRCP FRCR, Principal Investigator — Guy's and St Thomas's NHS Foundation Trust, London, UK
Locations (11):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Melbourne
  - Research Site, Melbourne, Parkville
  - Research Site, Randwick
- Research Site, Cologne, Germany
- Research Site, Hospitalet deLlobregat, Spain
- Research Site, Lund, Sweden

REFERENCES:
- [Derived] Matulonis UA, Penson RT, Domchek SM, Kaufman B, Shapira-Frommer R, Audeh MW, Kaye S, Molife LR, Gelmon KA, Robertson JD, Mann H, Ho TW, Coleman RL. Olaparib monotherapy in patients with advanced relapsed ovarian cancer and a germline BRCA1/2 mutation: a multistudy analysis of response rates and safety. Ann Oncol. 2016 Jun;27(6):1013-1019. doi: 10.1093/annonc/mdw133. Epub 2016 Mar 8. PMID 26961146
- [Derived] Ang JE, Gourley C, Powell CB, High H, Shapira-Frommer R, Castonguay V, De Greve J, Atkinson T, Yap TA, Sandhu S, Banerjee S, Chen LM, Friedlander ML, Kaufman B, Oza AM, Matulonis U, Barber LJ, Kozarewa I, Fenwick K, Assiotis I, Campbell J, Chen L, de Bono JS, Gore ME, Lord CJ, Ashworth A, Kaye SB. Efficacy of chemotherapy in BRCA1/2 mutation carrier ovarian cancer in the setting of PARP inhibitor resistance: a multi-institutional study. Clin Cancer Res. 2013 Oct 1;19(19):5485-93. doi: 10.1158/1078-0432.CCR-13-1262. Epub 2013 Aug 6. PMID 23922302
- [Derived] Audeh MW, Carmichael J, Penson RT, Friedlander M, Powell B, Bell-McGuinn KM, Scott C, Weitzel JN, Oaknin A, Loman N, Lu K, Schmutzler RK, Matulonis U, Wickens M, Tutt A. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and recurrent ovarian cancer: a proof-of-concept trial. Lancet. 2010 Jul 24;376(9737):245-51. doi: 10.1016/S0140-6736(10)60893-8. Epub 2010 Jul 6. PMID 20609468
- See also: CSR_Synopsis_D0810C00009(KU36-58).pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=734&filename=CSR_Synopsis_D0810C00009(KU36-58).pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on June 11, 2007 and efficacy and safety data were collected up to the data cut-off of March 17, 2009. Patients were enrolled at 12 centres in 5 countries: Australia, Germany, Spain, Sweden and the USA.
Pre-assignment Details: Two cohorts of women with Breast Cancer gene 1 (BRCA1)- or BRCA2-associated ovarian cancer who had failed at least one prior chemotherapy in the advanced/metastatic setting, were planned to receive olaparib 100 mg bd (n= up to 24) or 400 mg bd (n= up to 40). Enrolment to 2 cohorts was sequential with the 400 mg bd cohort being recruited first.
Groups:
- Olaparib 100 mg bd: olaparib (KU-0059436; AZD2281) 100 mg oral capsules, twice daily
- Olaparib 400 mg bd: olaparib (KU-0059436; AZD2281) 400 mg oral capsules, twice daily
Period: Overall Study
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd
Started | 24 (Patients received treatment) | 33 (Patients received treatment)
Completed | 7 (Patients completed the full study schedule (168 days treatment)) | 17 (Patients completed the full study schedule (168 days treatment))
Not Completed | 17 | 16
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 16 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Non-compliance | 0 | 1
Not completed — Intercurrent illness | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd | Total
Number analyzed (Participants) | 24 | 33 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (8.02) | 56.8 (10.49) | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 33 | 57
  Male | 0 | 0 | 0
BRCA mutation [Count of Participants; unit: Participants] — BRCA1 or BRCA2 mutations known to cause loss of gene function (clinical deleterious or suspected deleterious mutations).
  Participants
    BRCA1 | 19 | 21 | 40
    BRCA2 | 5 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Tumour Response (According to Response Evaluation Criteria In Solid Tumors (RECIST)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease from baseline in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Baseline, every 8 also at study termination or initiation of confounding anti-cancer therapy.
Population: PP Analysis Set (includes all enrolled patients who complete the trial schedule and medication regime without any major deviations to the protocol - this is the main analysis population, with ITT used to confirm)
Measure: Number; unit: Participants
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd
Number analyzed (Participants) | 24 | 33
Participants
  PP Analysis Set: number analyzed (Participants) | 22 | 31
  PP Analysis Set | 3 | 11
  ITT Analysis Set | 3 | 11

2. Secondary Outcome: Clinical Benefit (CB)
Description: Clinical Benefit (CB) is defined as the percentage of patients with a RECIST tumour response of confirmed complete response, partial response or stable disease for ≥8 weeks)
Time Frame: End of study
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd
Number analyzed (Participants) | 24 | 33
Percentage of participants | 45.5 [26.9 to 65.3] | 71.0 [53.4 to 83.9]

3. Secondary Outcome: Duration of Response
Description: Duration of response to olaparib
Time Frame: End of study
Population: PP Analysis Set (includes all enrolled patients who complete the trial schedule and medication regime without any major deviations to the protocol - this is the main analysis population, with ITT used to confirm
Measure: Median (Full Range); unit: Days
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd
Number analyzed (Participants) | 24 | 33
Days | 242 [169 to 288] | 301 [126 to 506]

4. Secondary Outcome: Best Percentage Change in Tumour Size
Description: The best % change (reduction) from baseline in tumour size (defined as the sum of the longest diameters as measured among all target lesions).
Time Frame: End of study
Population: as for outcome 3
Measure: Median (Full Range); unit: Percent change
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd
Number analyzed (Participants) | 24 | 33
Percent change | -5.1 [-85.7 to 66.1] | -25.8 [-100.0 to 150.0]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from first dose to the earlier date of radiologic progression (as per RECIST criteria) or death by any cause in the absence of objective progression.
Time Frame: End of study
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd
Number analyzed (Participants) | 24 | 33
Days | 62.5 [56 to 113] | 226 [105 to 338]

ADVERSE EVENTS:
Time Frame: From baseline, every visit until 30 days after last dose.
Arm/Group | Olaparib 100 mg bd | Olaparib 400 mg bd
All-Cause Mortality (participants affected / at risk) | 10/24 | 11/33
Serious Adverse Events (participants affected / at risk) | 7/24 | 12/33
Other Adverse Events (participants affected / at risk) | 23/24 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib 100 mg bd (N=24) | Olaparib 400 mg bd (N=33)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood Pressure Increased (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib 100 mg bd (N=24) | Olaparib 400 mg bd (N=33)
Anaemia (Blood and lymphatic system disorders) | 3 | 7
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 15 | 21
Diarrhoea (Gastrointestinal disorders) | 7 | 12
Abdominal Pain (Gastrointestinal disorders) | 4 | 9
Vomiting (Gastrointestinal disorders) | 6 | 11
Constipation (Gastrointestinal disorders) | 6 | 4
Abdominal Distension (Gastrointestinal disorders) | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 3
Gastrointestinal Pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 13 | 17
Oedema Peripheral (General disorders) | 1 | 6
Pyrexia (General disorders) | 2 | 2
Asthenia (General disorders) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 5 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3
Oral Herpes (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2
Herpes Zoster (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 4
Waist Circumference Increased (Investigations) | 4 | 0
Haemoglobin Urine (Investigations) | 3 | 0
Blood Urine Present (Investigations) | 2 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 7
Neuropathy Peripheral (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 3
Dysgeusia (Nervous system disorders) | 2 | 1
Sinus Headache (Nervous system disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 2
Pollakiuria (Renal and urinary disorders) | 2 | 0
Pelvic Pain (Reproductive system and breast disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review and comment prior to publication. In order to ensure that the Sponsor will be able to make comments and suggestions where pertinent, material for public dissemination will be submittted to the Sponsor for review at least sixty (60) days prior to submission for publication, public dissemination, or review by a publication committee